CLINICAL TRIAL: NCT02017704
Title: Chemoradiation OR Brachytherapy for RECTal Cancer
Acronym: CORRECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Elekta Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: J1360; NA_00082167 (Other: JHMIRB)
Record Dates: First submitted 2013-12-05; First posted 2013-12-23 (Estimated); Results first posted 2023-02-24 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Rectal Cancer
Keywords: Endorectal Brachytherapy Radiation Therapy; Intensity Modulated Radiation Therapy and Capecitabine
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Radiotherapy, Intensity-Modulated; Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- IMRT and Capecitabine (Active Comparator): Patients will receive IMRT along with capecitabine. External radiotherapy will be based on contouring guidelines from the RTOG atlas and Radiation Therapy Oncology Group (RTOG 0822) with some modifications
  Followed by:
  * Oxaliplatin: 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * 5-Fluorouracil (5-FU) bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5-FU continuous infusion 2400 mg/m², 46-h infusion following the 5-FU bolus
  Cycle length: 14 days (2 weeks)
  Duration of treatment: 12 cycles
  Then: Surgical Resection
  Interventions: Drug: capecitabine and IMRT (if randomized to this arm); Radiation: IMRT (intensity modulated radiation therapy); Drug: FOLFOX6; Procedure: Surgery
- Endo-HDR (Experimental): Patients will be treated with a daily dose of 6.5 Gy over four consecutive days for a total of 26 Gy
  Followed by:
  * Oxaliplatin: 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * 5-Fluorouracil (5-FU) bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5-FU continuous infusion 2400 mg/m², 46-h infusion following the 5-FU bolus
  Cycle length: 14 days (2 weeks)
  Duration of treatment: 12 cycles
  Then: Surgical Resection
  Interventions: Radiation: Endo-HDR (if randomized to this arm); Drug: FOLFOX6; Procedure: Surgery

INTERVENTIONS:
Radiation: Endo-HDR (if randomized to this arm) — Patients will be treated with a daily dose of 6.5 Gy over four consecutive days for a total of 26 Gy
  Arms: Endo-HDR
Drug: capecitabine and IMRT (if randomized to this arm) — Capecitabine shall be delivered at 825mg/m2 BID during IMRT radiotherapy
  Other Names: Xeloda
  Arms: IMRT and Capecitabine
Radiation: IMRT (intensity modulated radiation therapy) — Patients will receive IMRT along with capecitabine. External radiotherapy will be based on contouring guidelines from the RTOG atlas and Radiation Therapy Oncology Group (RTOG 0822) with some modifications
  Arms: IMRT and Capecitabine
Drug: FOLFOX6 — * Oxaliplatin - 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * Leucovorin - bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5 Fluorouracil (5FU) - 2400 mg/m², 46-h infusion following the 5-FU bolus An outpatient, 46 hour continuous IV infusion provided by a home IV infusion company. The 5FU is delivered by a small pump worn in a fanny pack around the waist. The home IV infusion company will arrange your disconnect at the end of the infusion.
  Other Names: Oxaliplatin, Leucovorin, 5 Fluorouracil
Procedure: Surgery — After the patient has been identified as a candidate for the trial, the surgeon will assess the patient and will determine:
  Exact height and location of tumor with regards to the anal margin as measured by a rigid or flexible proctoscope and/or digital exam.
  Mobility of tumor as assessed if possible by rectal exam Type of surgical procedure: Abdominoperineal resection vs. sphincter saving procedures, which will include colo-anal with mucosectomy vs. stapled anastomosis.

SUMMARY:
This research is being done to compare the effectiveness of high dose endorectal brachytherapy (END-HDR) and the standard treatment option of chemoradiation with Capecitabine in the treatment of cancer of the lowest part of the bowel (rectum).

DETAILED DESCRIPTION:
Locally advanced rectal carcinoma continues to be a major oncologic problem in the United States with approximately 40,000 new cases diagnosed in 2011. For stage II/III rectal carcinoma, adjuvant chemoradiation and total mesorectal excision (TME) represent the major treatment advances that have increased cure rates over the past 30 years.

In the setting of TME, a landmark phase III German trial of stage II/III rectal cancer patients established neoadjuvant 5FU-based chemoradiation (NCRT) as standard of care over the same regimen given post-operatively. The preoperative arm showed superior local control (6% vs. 13% p=0.006), a complete pathologic response of 8%, a higher rate of sphincter preservation and less grade 3 toxicity compared to post-operative treatment. However, disease-free and overall survival (76% versus 74%, respectively) were no different because of the high rate of distant metastasis occurring in over 1/3 of patients (5yr DM 36 vs 38%,p=0.84). Importantly, those attaining a pathologic complete response had a decreased rate of distant metastasis and improved disease-free survival. Drawbacks to the regimen include acute grade 3 or 4 toxicity in 27% of patients, low compliance rates with postoperative chemotherapy (27 - 50%), and an overall decline in anorectal function shown by long-term studies.

Given the excellent locoregional control reported in TME surgical series, several trials have investigated whether certain patients may be spared preoperative radiotherapy. Two large randomized trials by Dutch and British investigators showed that a short preoperative course of hypofractionated EBRT (25 Gy in 5 fractions) followed by TME surgery decreased locoregional recurrence by 2/3 as compared to patients treated with TME surgery alone. In the Dutch trial, patients with mid and distal rectal cancers were most likely to benefit from radiotherapy. In these patients, preoperative radiation was shown to decrease locoregional recurrence by 5-fold (10% to 2%); however, the hypofractionated preoperative EBRT regimen was associated with a significant increase in acute and chronic morbidity. Indeed, the Dutch study revealed that irradiated patients, when compared to surgery alone, had more perineal wound healing problems after abdominoperineal resection (29% vs. 19%), worsening deterioration of anal sphincter dysfunction, and more severe long-term effects related to sexual functioning both in males (p=0.004) and females (p<0.002). Additionally, colleagues have reported a consistent negative impact on bowel function in those patients undergoing sphincter preservation. In reviewing the long-term data of the Swedish short course preoperative EBRT rectal cancer trial, Birgisson also reported a higher incidence of secondary tumors (9.5%) in patients treated with preoperative radiation when compared to patients having surgery alone (4.3%).

Modern approaches to address the risk of distant metastasis and poor compliance with adjuvant systemic chemotherapy (following NCRT) have incorporated newer effective chemotherapy agents earlier in the treatment protocol. For example, oxaliplatin has been one of the most widely studied agents as a result of its proven efficacy when combined with 5-fluorouracil and leucovorin (FOLFOX) both in the metastatic and adjuvant settings for colon cancer. Initial phase II studies with the addition of oxaliplatin to standard 5-FU based NCRT appeared to show improved pathologic complete response rates compared to standard NCRT. However, two phase III trials clearly show that the addition of oxaliplatin during 5FU-based NCRT does not significantly improve pathologic complete response, locoregional control, distant metastasis or survival but does increase acute grade 3-4 toxicity by two to three-fold.

One approach to limit toxicity from external beam radiotherapy is the use of intensity modulated radiation therapy (IMRT). IMRT can limit radiation dose to normal rectum (above and below the tumor) and surrounding organs at risk (OARs) such as bladder and sexual organs. IMRT utilizes multiple beams of radiation to treat the rectal tumor plus a margin and limits dose to OARs. While IMRT decreases radiation dose to normal structures, it requires an additional 2-3 cm margin for microscopic extension (clinical treatment volume=CTV), set-up error, and rectal motion (planning treatment volume=PTV). Furthermore, IMRT still requires 5-6 weeks of radiation with concurrent chemotherapy, is substantially more expensive than conformal radiation, and is especially prohibitive in countries where access to technology necessary for IMRT is limited. Based on the preliminary results of RTOG 0822 and others, it still remains to be determined whether IMRT confers a statistically significant improvement in pCR, toxicity rates and QOL relative to standard NCRT.

A novel approach to limit radiation toxicity is the use of high dose rate endorectal brachytherapy (Endo-HDR). Endo-HDR involves the placement of a silicon multicatheter applicator within the rectum to deliver large doses to the rectal tumor and mesorectum with rapid dose fall off to the surrounding organs. An Iridium 192 high dose rate brachytherapy source attached to a wire is inserted into each catheter to deliver a high dose of radiation therapy the tumor. High dose rate brachytherapy has been well established in various malignancies (prostate, uterine, sarcoma, head and neck) to escalate radiation dose to the tumor over a short period of time while sparing normal tissue. Compared with NCRT and IMRT, Endo-HDR delivers treatment internally to the tumor without having to pass through surrounding normal tissue and organs. It requires smaller margins (CTV/PTV=~1 cm) on the tumor since the applicator is positioned under fiducial guidance over the tumor without need for a margin for organ motion allowing greater sparing of OARs. Furthermore, the area of the rectum exposed to high dose radiotherapy is surgically removed at the time of resection which further minimizes chronic toxicity. Important structures that may be spared include bone marrow, small bowel, bladder, the autonomic nerves, sexual organs, anal sphincter and skin. Considering that 1/3 of patients will develop metastases, limiting bone marrow toxicity may contribute to better compliance with systemic treatment and allow for a better treatment strategy to target systemic recurrence. Another distinct advantage of Endo-HDR is the shortened treatment time (1 versus 6 weeks). Endo-HDR therefore provides a major logistic advantage for patients who may benefit from neoadjuvant therapy but who are geographically distant from radiation centers, elderly, or medically infirmed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed adenocarcinoma of the rectum
* Appropriate tumor staging and location
* Patients should be suitable candidates for surgery and chemotherapy
* ECOG/WHO performance status 0-1
* Patients must be 18 years or older
* No previous history of pelvic radiation
* Patients must have acceptable organ and marrow function
* Non pregnant, non-breast feeding females under active contraception
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Evidence of distant metastatic disease
* Evidence of sphincter invasion on MRI
* Prior history of radiation to the pelvis
* Prior malignancy except for adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ, DCIS, or other cancer from which the patient has been disease free for at least 3 years
* Presence of multiple small bowel loops trapped within the immediate tumor bed (post hysterectomy or prostatectomy).
* Use of any investigational agent within the 4 weeks preceding enrollment
* Previous exposure to chemotherapy for rectal cancer
* Uncontrolled intercurrent illness including but not limited to, ongoing or active infections (or infections requiring systemic treatment), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and breastfeeding women are excluded, as well as women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control (hormonal or barrier method of birth control; abstinence) to avoid pregnancy for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study she should inform her treating physician immediately.
* Women who are not post-menopausal and have a positive urine or serum pregnancy test or refuse to take a pregnancy test.
* Contraindication for safe MRI, implants, or other conditions that interfere with imaging required for the study (e.g., pacemaker or non-MRI compatible hip prostheses). Note: Subjects with bilateral hip implants are not eligible for the study. Subjects with a unilateral hip implant may be eligible assuming the implant is MRI compatible and does not present artifact on MRI in the areas of interest.
* Subject is pacemaker dependent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amol K Narang, M.D., Principal Investigator — The SKCCC at Johns Hopkins
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - The SKCCC at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IMRT and Capecitabine: Patients will receive IMRT along with capecitabine.
  Followed by:
  * Oxaliplatin: 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * 5-Fluorouracil (5-FU) bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5-FU continuous infusion 2400 mg/m², 46-h infusion following the 5-FU bolus Cycle length: 14 days (2 weeks); Duration of treatment: 12 cycles
  Then: Surgical Resection
  capecitabine and IMRT (if randomized to this arm): Capecitabine shall be delivered at 825mg/m2 BID during IMRT radiotherapy
  IMRT (intensity modulated radiation therapy): Patients will receive IMRT along with capecitabine.
  External radiotherapy will be based on contouring guidelines from the RTOG atlas and Radiation Therapy Oncology Group (RTOG 0822) with some modifications
  FOLFOX6: * Oxaliplatin - 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * Leucovorin - bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5 Fluorouracil (5FU) - 2400 mg/m², 46-h infusion following the 5-FU bolus
  Surgery: After the patient has been identified as a candidate for the trial, the surgeon will assess the patient and will determine:
  Exact height and location of tumor with regards to the anal margin as measured by a rigid or flexible proctoscope and/or digital exam.
  Mobility of tumor as assessed if possible by rectal exam Type of surgical procedure: Abdominoperineal resection vs. sphincter saving procedures, which will include colo-anal with mucosectomy vs. stapled anastomosis.
- Endo-HDR: Patients will be treated with a daily dose of 6.5 Gy over four consecutive days for a total of 26 Gy
  Followed by:
  * Oxaliplatin: 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * 5-Fluorouracil (5-FU) bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5-FU continuous infusion 2400 mg/m², 46-h infusion following the 5-FU bolus Cycle length: 14 days (2 weeks); Duration of treatment: 12 cycles
  Then: Surgical Resection
  Endo-HDR (if randomized to this arm): Patients will be treated with a daily dose of 6.5 Gy over four consecutive days for a total of 26 Gy
  FOLFOX6: * Oxaliplatin - 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * Leucovorin - bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5 Fluorouracil (5FU) - 2400 mg/m², 46-h infusion following the 5-FU bolus
  Surgery: After the patient has been identified as a candidate for the trial, the surgeon will assess the patient and will determine: Exact height and location of tumor with regards to the anal margin as measured by a rigid or flexible proctoscope and/or digital exam.; Mobility of tumor as assessed if possible by rectal exam; Type of surgical procedure: Abdominoperineal resection vs. sphincter saving procedures, which will include colo-anal with mucosectomy vs. stapled anastomosis.
Period: Overall Study
Arm/Group | IMRT and Capecitabine | Endo-HDR
Started | 4 | 5
Completed | 2 | 5
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMRT and Capecitabine | Endo-HDR | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white/caucasian | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 5 | 9
met baseline enrollment requirements as per protocol [Count of Participants; unit: Participants] | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pathologic Complete Response
Description: Pathologic complete response rate is reported as the number of patients who achieve pathologic complete response after the treatment for each arm.
  As per the NCCN guidelines, pathologic response is graded by the system recommended by the AJCC Cancer Staging Manual and CAP guidelines:
  * Complete response - no remaining viable cancer cells
  * Moderate response - only small clusters/single cancer cells remain
  * Minimal response - residual cancer remaining, but with predominant fibrosis
  * Poor response - minimal/no tumor kills, extensive residual cancer
Time Frame: Up to 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT and Capecitabine | Endo-HDR
Number analyzed (Participants) | 2 | 5
Participants | 0 | 2

2. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: Number of participants with grade 3 or higher adverse events will be listed by relationship.
  Grading is by CTCAE 4 guidelines.
  Relationship, as determined by PI, is unrelated/unlikely/possible/probable/definite.
Time Frame: Up to 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT and Capecitabine | Endo-HDR
Number analyzed (Participants) | 2 | 5
Participants
  Grade: 3; Relationship: probable | 1 | 1
  Grade: 3; Relationship: possible | 1 | 1
  Grade 3; Relationship: Unlikely | 1 | 0

3. Secondary Outcome: Change in EORTC QLQ-C30 Global Health Status Score
Description: Patients were given the EORTC QLQ-C30 at baseline, preop, postop, and at follow ups Y1-5. The forms were scored as per the manual available at EORTC. Raw scores are transformed to fall in a range of 0-100. Generally, higher scores on QoL scales represent higher levels of QoL.
  The scores are reported as the mean of the Global Health Status/QoL scale score when more than 1 patient completed the form for a time point. If only 1 form was available for a time point, then the score for that form is reported.
Time Frame: baseline, preop, postop, and at follow ups Y1-5
Population: 3 patients randomised to IMRT arm had at least 1 form completed. 5 patients randomised to the ENDO arm had at least 1 form completed.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | IMRT and Capecitabine | Endo-HDR
Number analyzed (Participants) | 3 | 5
score on a scale
  baseline: number analyzed (Participants) | 2 | 5
  baseline | 83 [83 to 83] | 71.2 [41 to 83]
  pre-op: number analyzed (Participants) | 1 | 5
  pre-op | 33 [33 to 33] | 49.6 [8 to 83]
  post-op: number analyzed (Participants) | 2 | 4
  post-op | 54 [33 to 75] | 72.5 [50 to 91]
  year 1: number analyzed (Participants) | 0 | 5
  year 1 |  | 73 [33 to 100]
  year 2: number analyzed (Participants) | 1 | 3
  year 2 | 50 [50 to 50] | 66.3 [33 to 83]
  year 3: number analyzed (Participants) | 2 | 3
  year 3 | 66.5 [50 to 83] | 77.3 [66 to 83]
  year 4: number analyzed (Participants) | 1 | 1
  year 4 | 83 [83 to 83] | 91 [91 to 91]
  year 5: number analyzed (Participants) | 0 | 2
  year 5 |  | 91.5 [83 to 100]

4. Secondary Outcome: Time to Death
Description: Assessing the difference time to death rates among study participants.
Time Frame: Up to 60 months
Population: No patients were deceased during the study period.
Groups:
- IMRT and Capecitabine (Potentially Randomized to This Arm): Patients will receive IMRT along with capecitabine.
  Followed by:
  * Oxaliplatin: 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * 5-Fluorouracil (5-FU) bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5-FU continuous infusion 2400 mg/m², 46-h infusion following the 5-FU bolus Cycle length: 14 days (2 weeks); Duration of treatment: 12 cycles
  Then: Surgical Resection
  capecitabine and IMRT (if randomized to this arm): Capecitabine shall be delivered at 825mg/m2 BID during IMRT radiotherapy
  IMRT (intensity modulated radiation therapy): Patients will receive IMRT along with capecitabine.
  External radiotherapy will be based on contouring guidelines from the RTOG atlas and Radiation Therapy Oncology Group (RTOG 0822) with some modifications
  FOLFOX6: * Oxaliplatin - 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * Leucovorin - bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5 Fluorouracil (5FU) - 2400 mg/m², 46-h infusion following the 5-FU bolus
  Surgery: After the patient has been identified as a candidate for the trial, the surgeon will assess the patient and will determine:
  Exact height and location of tumor with regards to the anal margin as measured by a rigid or flexible proctoscope and/or digital exam.
  Mobility of tumor as assessed if possible by rectal exam Type of surgical procedure: Abdominoperineal resection vs. sphincter saving procedures, which will include colo-anal with mucosectomy vs. stapled anastomosis.
- Endo-HDR (Potentially Randomized to This Arm): Patients will be treated with a daily dose of 6.5 Gy over four consecutive days for a total of 26 Gy
  Followed by:
  * Oxaliplatin: 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * 5-Fluorouracil (5-FU) bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5-FU continuous infusion 2400 mg/m², 46-h infusion following the 5-FU bolus Cycle length: 14 days (2 weeks); Duration of treatment: 12 cycles
  Then: Surgical Resection
  Endo-HDR (if randomized to this arm): Patients will be treated with a daily dose of 6.5 Gy over four consecutive days for a total of 26 Gy
  FOLFOX6: * Oxaliplatin - 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * Leucovorin - bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5 Fluorouracil (5FU) - 2400 mg/m², 46-h infusion following the 5-FU bolus
  Surgery: After the patient has been identified as a candidate for the trial, the surgeon will assess the patient and will determine: Exact height and location of tumor with regards to the anal margin as measured by a rigid or flexible proctoscope and/or digital exam.; Mobility of tumor as assessed if possible by rectal exam; Type of surgical procedure: Abdominoperineal resection vs. sphincter saving procedures, which will include colo-anal with mucosectomy vs. stapled anastomosis.
Arm/Group | IMRT and Capecitabine (Potentially Randomized to This Arm) | Endo-HDR (Potentially Randomized to This Arm)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Distant Metastases Free Survival
Description: Compare distant metastasis for both Endo-HDR and CRT.
Time Frame: Up to 60 months
Population: No patients had metastases during study period.
Arm/Group | IMRT and Capecitabine (Potentially Randomized to This Arm) | Endo-HDR (Potentially Randomized to This Arm)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Progression Free Survival
Description: Compare progression free survival for both Endo-HDR and CRT.
Time Frame: Up to 60 months
Population: No patients had progression during study period.
Arm/Group | IMRT and Capecitabine (Potentially Randomized to This Arm) | Endo-HDR (Potentially Randomized to This Arm)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Local Disease Recurrence
Description: Compare locoregional control for both Endo-HDR and CRT.
Time Frame: Up to 60 months
Population: No patients had locoregional recurrence during study period.
Arm/Group | IMRT and Capecitabine (Potentially Randomized to This Arm) | Endo-HDR (Potentially Randomized to This Arm)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 months
Groups:
- IMRT and Capecitabine: Patients will receive IMRT along with capecitabine.
  Followed by:
  * Oxaliplatin: 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * 5-Fluorouracil (5-FU) bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5-FU continuous infusion 2400 mg/m², 46-h infusion following the 5-FU bolus Cycle length: 14 days (2 weeks); Duration of treatment: 12 cycles
  Then: Surgical Resection capecitabine and IMRT (if randomized to this arm): Capecitabine shall be delivered at 825mg/m2 BID during IMRT radiotherapy
  IMRT (intensity modulated radiation therapy): Patients will receive IMRT along with capecitabine.
  External radiotherapy will be based on contouring guidelines from the RTOG atlas and Radiation Therapy Oncology Group (RTOG 0822) with some modifications
  FOLFOX6: * Oxaliplatin - 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * Leucovorin - bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5 Fluorouracil (5FU) - 2400 mg/m², 46-h infusion following the 5-FU bolus
  Surgery: After the patient has been identified as a candidate for the trial, the surgeon will assess the patient and will determine: Exact height and location of tumor with regards to the anal margin as measured by a rigid or flexible proctoscope and/or digital exam; Mobility of tumor as assessed if possible by rectal exam; Type of surgical procedure: Abdominoperineal resection vs. sphincter saving procedures, which will include colo-anal with mucosectomy vs. stapled anastomosis.
- Endo-HDR: Patients will be treated with a daily dose of 6.5 Gy over four consecutive days for a total of 26 Gy
  Followed by:
  * Oxaliplatin: 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * 5-Fluorouracil (5-FU) bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5-FU continuous infusion 2400 mg/m², 46-h infusion following the 5-FU bolus Cycle length: 14 days (2 weeks); Duration of treatment: 12 cycles
  Then: Surgical Resection:
  Endo-HDR: Patients will be treated with a daily dose of 6.5 Gy over four consecutive days for a total of 26 Gy
  FOLFOX6: * Oxaliplatin - 85 mg/m² in 500ml glucose 5% solution, 2-h infusion
  * Leucovorin - bolus 400mg/m² following the oxaliplatin/FA infusions
  * 5 Fluorouracil (5FU) - 2400 mg/m², 46-h infusion following the 5-FU bolus;
  Surgery: After the patient has been identified as a candidate for the trial, the surgeon will assess the patient and will determine: Exact height and location of tumor with regards to the anal margin as measured by a rigid or flexible proctoscope and/or digital exam; Mobility of tumor as assessed if possible by rectal exam; Type of surgical procedure: Abdominoperineal resection vs. sphincter saving procedures, which will include colo-anal with mucosectomy vs. stapled anastomosis.
Arm/Group | IMRT and Capecitabine | Endo-HDR
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT and Capecitabine (N=4) | Endo-HDR (N=5)
anemia (Blood and lymphatic system disorders) | 1 | 0 — Grade 3
proctitis (Gastrointestinal disorders) | 1 | 0 — Grade 3
sacral decubitis ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 — Grade 3
fatigue (General disorders) | 0 | 1 — Grade 3
pain (NOS) (General disorders) | 0 | 1 — Grade 3
rectovaginal fistula (Reproductive system and breast disorders) | 0 | 1 — Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT and Capecitabine (N=4) | Endo-HDR (N=5)
ANC elevated (Investigations) | 1 | 0 — Grade not specified
alanine amino transferase increased (Investigations) | 0 | 2 — Grade 1
anemia (Blood and lymphatic system disorders) | 1 | 3 — Grade 1
aspartate amino transferase increased (Investigations) | 0 | 1 — Grade 1
bilirubin increased (Investigations) | 1 | 0 — Grade 1
constipation (Gastrointestinal disorders) | 2 | 3 — Grade 1
creatinine decreased (Investigations) | 1 | 0 — Grade 1
creatinine increased (Investigations) | 1 | 0 — Grade 1
dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 — Grade 1
diarrhea (Gastrointestinal disorders) | 2 | 3 — Grade 1
dyspareunia (Reproductive system and breast disorders) | 1 | 0 — Grade 1
dyspepsia (Gastrointestinal disorders) | 1 | 1 — Grade 1
fatigue (General disorders) | 1 | 3 — Grade 1
fecal incontinence (Gastrointestinal disorders) | 1 | 0 — Grade 1
GI hemorrhage (Gastrointestinal disorders) | 1 | 4 — Grade 1
hematuria (Renal and urinary disorders) | 1 | 0 — Grade 1
hemorrhoids (Gastrointestinal disorders) | 2 | 1 — Grade 1
hyperglycemia (Metabolism and nutrition disorders) | 2 | 3 — Grade 1
hypokalemia (Metabolism and nutrition disorders) | 1 | 0 — Grade 1
hyponatremia (Metabolism and nutrition disorders) | 1 | 0 — Grade 1
lymphocytes decreased (Investigations) | 2 | 0 — Grade 1
nausea (Gastrointestinal disorders) | 3 | 4 — Grade 1
nocturia (Renal and urinary disorders) | 2 | 4 — Grade 1
pain (NOS) (General disorders) | 2 | 2 — Grade 1
proctitis (Gastrointestinal disorders) | 2 | 1 — Grade 1
rectal pain (Gastrointestinal disorders) | 2 | 3 — Grade 1
urinary frequency/urgency (Renal and urinary disorders) | 2 | 2 — Grade 1
urinary retention (Renal and urinary disorders) | 2 | 0 — Grade 1
WBC decreased (Investigations) | 1 | 1 — Grade 1
anorexia (Investigations) | 0 | 1 — Grade 2
atrial flutter (Cardiac disorders) | 0 | 1 — Grade 2
constipation (Gastrointestinal disorders) | 0 | 1 — Grade 2
diarrhea (Gastrointestinal disorders) | 0 | 1 — Grade 2
dyspareunia (Reproductive system and breast disorders) | 1 | 0 — Grade 2
erectile dysfunction (Reproductive system and breast disorders) | 2 | 1 — Grade 2
fatigue (General disorders) | 1 | 0 — Grade 2
GI hemorrhage (Gastrointestinal disorders) | 0 | 1 — Grade 2
hemorrhoids (Gastrointestinal disorders) | 2 | 0 — Grade 2
hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 — Grade 2
hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 — Grade 2
lymphocytes decreased (Investigations) | 1 | 0 — Grade 2
nausea (Gastrointestinal disorders) | 0 | 1 — Grade 2
nocturia (Renal and urinary disorders) | 1 | 0 — Grade 2
pain (NOS) (General disorders) | 1 | 1 — Grade 2
peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 — Grade 2
proctitis (Gastrointestinal disorders) | 0 | 2 — Grade 2
rectal bleeding (Gastrointestinal disorders) | 0 | 1 — Grade 2
rectal pain (Gastrointestinal disorders) | 1 | 1 — Grade 2
rectal stenosis (Gastrointestinal disorders) | 0 | 1 — Grade 2
urinary frequency/urgency (Renal and urinary disorders) | 1 | 0 — Grade 2
vaginal discharge (Reproductive system and breast disorders) | 0 | 1 — Grade 2
vaginal dryness (Reproductive system and breast disorders) | 1 | 0 — Grade 2
vaginal pain (Reproductive system and breast disorders) | 1 | 0 — Grade 2
vomiting (Gastrointestinal disorders) | 0 | 1 — Grade 2
WBC decreased (Investigations) | 1 | 0 — Grade 2
weight loss (Investigations) | 0 | 1 — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT02017704/Prot_SAP_000.pdf